CLINICAL TRIAL: NCT00863837
Title: Prevention of Esophageal Variceal Rebleeding
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Gin-Ho Lo, Kaohsiung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSC
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Esophageal Variceal Rebleeding
Keywords: Acute variceal bleeding; banding ligation; vasoconstrictor; proton pump inhibitor
MeSH Terms: interventions — Terlipressin; Vasoconstrictor Agents; Proton Pump Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): add pantoloc to reduce ulcer bleeding after banding ligation
  Interventions: Drug: pantoloc (proton pump inhibitor)
- Arm B: ligation + terlipressin 1mg q6h (Placebo Comparator): Arm B, intervention: ligation + terlipressin 1mg q6h
  Interventions: Drug: terlipressin (vasoconstrictor)

INTERVENTIONS:
Drug: terlipressin (vasoconstrictor) — Ligation plus terlipressin 1mg q6h
  Other Names: vasoconstrictor
  Arms: Arm B: ligation + terlipressin 1mg q6h
Drug: pantoloc (proton pump inhibitor) — Pantoloc infusion (1 vial q.d.); Using pantoloc to reduce rebleed after EVL
  Other Names: proton pump inhibitor
  Arms: Arm A

SUMMARY:
BACKGROUND: Previous studies showed that the combination of endoscopic therapy with vasoconstrictor is better than either vasoconstrictor or endoscopic therapy alone in achieving the successful hemostatsis of acute variceal bleeding. The rationale of using vasoconstrictor is to enhance the efficacy of hemostasis by endoscopic therapy. Nowadays, endoscopic variceal ligation (EVL) has replaced endoscopic injection sclerotherapy (EIS) as the endoscopic treatment of choice in the arresting of acute esophageal variceal hemorrhage. EVL alone can achieve hemotasis up to 97% even in cases of active variceal hemorrhage. However, early rebleeding due to ligation-induced ulcer may be encountered. It appears that prevention of esophageal ulcers and bleeding by a proton pump inhibitor may be more logical than using a vasoconstrictor after cessation of bleeding by EVL.

Thus, the investigators designed a controlled trial to compare the initial hemostasis, early rebleeding rate in cirrhotic patients presenting with acute variceal bleeding receiving either emergency EVL plus vasoconstrictor infusion or losec infusion for 5 days.

DETAILED DESCRIPTION:
Methods of treatment:

Group 1: Somatostatin 250μg slow bolus IV infusion followed by 250μg per hour (6mg/ 24 hours) or Terlipressin 2mg bolus was instituted on enrollment followed by 1mg per 6 hours for 5 days. The use of either somatostatin or glypressin was at the discretion of doctors in charge. Group 2: Pantoloc 20 mg intravenously per day was instituted on enrollment and continued for 5 days.

Definition of initial hemostasis:

Initial hemostasis was defined as achieving a 24h bleeding-free period within the first 48h after treatment together with stable vital signs based on Baveno consensus criteria.

Very early rebleeding was defined as: UGI bleeding occurred after initial hemostasis and within 5 days after enrollment. UGI bleeding was proven to be from esophageal varices.

Treatment failure is defined as failure to control acute bleeding episodes or very early rebleeding.

ELIGIBILITY:
Inclusion Criteria:

1. The etiology of portal hypertension is cirrhosis.
2. Age ranges between 18-80 y/o.
3. Patients presenting with acute esophageal variceal bleeding proven by emergency endoscopy within 12 hours. (Acute esophageal variceal bleeding was defined as:

   * when blood was directly seen by endoscopy to issue from an esophageal varix (active bleeding) OR
   * when patients presented with red color signs on their esophageal varices with blood in esophagus or stomach and no other potential site of bleeding identified (inactive bleeding).
4. EVL is performed after confirmation of acute esophageal variceal bleeding. Enrollment time: Immediately after EVL is completed and variceal bleeding is arrested.

Exclusion criteria:

1. association with severe systemic illness, such as sepsis, COPD, uremia
2. association with gastric variceal bleeding
3. failure in the control of bleeding by emergency EVL
4. moribund patients, died within 12 hours of enrollment
5. Uncooperative
6. Ever received EIS, EVL within one month prior to index bleeding
7. Child-Pugh's scores > 10

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-12; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
very early rebleeding | 5 days

SECONDARY OUTCOMES:
mortality, complications | 42 days